CLINICAL TRIAL: NCT06007664
Title: Leveraging Social Networks: a Novel Physical Activity Intervention for Senior Housing
Brief Title: Tele-video to Improve Daily Activity
Acronym: T-VIDA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Noah J Webster, Associate Research Scientist, Survey Research Center, Institute for Social Research, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: HUM00224610; 1K01AG062754-01A1 (NIH)
Record Dates: First submitted 2023-08-17; First posted 2023-08-23 (Actual); Results first posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Physical Inactivity
Keywords: physical activity; physical function
MeSH Terms: conditions — Sedentary Behavior; Motor Activity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- occupational therapy intervention group (Experimental)
  Interventions: Behavioral: Tele-Video to Improve Daily Activity

INTERVENTIONS:
Behavioral: Tele-Video to Improve Daily Activity — Participants will be asked to meet individually with an Occupational Therapist (OT) via Zoom to assess activity performance, establish short-term activity goals, and outline an individualized home exercise program. Participants will also be asked to participate in 4 weekly one hour group sessions via Zoom that will include: 1) education; 2) OT facilitated discussion; and 3) activity demonstration, engagement and feedback. The following topics will be covered: mobility, physical activity, pain management, and energy conservation. Participants will be asked to meet individually with the OT via Zoom for 15-20 minutes weekly to answer questions. At the end, participants will be asked to again meet individually with the OT via Zoom to re-assess activity performance and revisit short-term activity goals and the individualized home exercise program. Advisory Committee Members will be asked to make note of intervention activities during their regular interactions with other participants.

SUMMARY:
This pilot study will test the feasibility of pairing a social network-based approach with a 6-week Occupational Therapist (OT)-led intervention administered remotely (via Zoom) to increase physical function and activity among residents of a HUD subsidized independent-living senior housing community. The intervention is called Tele-Video to Improve Daily Activity (T-VIDA) and will be administered with two cohorts of residents in a single community. The study has two main goals: 1) To determine if an OT-led program administered remotely over the internet using Zoom is useful in helping residents increase their physical activity; and 2) to determine if involving respected members of the community in the program as Advisory Committee members has an impact on how much other residents participate in program activities and engage in behaviors discussed. The OT intervention will be comprised of a combination of adapted components from multiple evidence-based interventions including individual meetings with an OT and OT-led group sessions. To evaluate the intervention pre- and post-program interviews will be conducted with participants over the phone, and activity monitoring will be conducted after both the pre- and post-program interviews for 7-days using an activity monitoring device. The following hypotheses will be tested: 1) at least 75% (3 of 4) of identified residents will accept the invitation to serve on the Advisory Committee; 2) Advisory Committee Members will attend at least 2 of 3 committee meetings; 3) Participants will on average participate in at least 70% (7 of 10) of intervention activities; 4) Residents knowing one or more committee members at baseline will participate in more intervention activities compared to those who do not; and 5) The influence of knowing a committee member on participation will be greater among residents reporting more pain at baseline compared to those reporting less pain.

ELIGIBILITY:
Inclusion Criteria:

* resident of the senior housing community of focus
* English-proficient
* ambulatory with or without assistive device (e.g., cane, walker)

Exclusion Criteria:

* requiring use of a wheelchair for ambulation;
* requiring highly specialized equipment (e.g., spinal cord injury, leg amputation, wound vacuum assisted closure, heavy leg boot);
* hospitalized within last 3 months;
* has probable dementia (TICSm score <27);
* requiring ongoing complicated treatments (e.g., home oxygen use >2 liters);
* has active mental health condition judged to pose significant barrier to participation; and
* meets CDC recommendations for physical activity (150+ minutes of moderate-intensity aerobic activity during typical week).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2023-08-23 (Actual); Primary Completion 2024-11-26 (Actual); Study Completion 2024-12-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Noah J Webster, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Starting 6 months after publication

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental: occupational therapy intervention group: Behavioral: Tele-Video to Improve Daily Activity Participants will be asked to meet individually with an Occupational Therapist (OT) via Zoom to assess activity performance, establish short-term activity goals, and outline an individualized home exercise program. Participants will also be asked to participate in 4 weekly one hour group sessions via Zoom that will include: 1) education; 2) OT facilitated discussion; and 3) activity demonstration, engagement and feedback. The following topics will be covered: mobility, physical activity, pain management, and energy conservation. Participants will be asked to meet individually with the OT via Zoom for 15-20 minutes weekly to answer questions. At the end, participants will be asked to again meet individually with the OT via Zoom to re-assess activity performance and revisit short-term activity goals and the individualized home exercise program. Advisory Committee Members will be asked to make note of intervention activities during their regular interactions with other participants. Advisory Committee Members will be selected from the group of enrolled participants, and will not be considered additional participants in the study.
Period: Overall Study
Arm/Group | Experimental: occupational therapy intervention group
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Experimental: Occupational Therapy Intervention Group
Number analyzed (Participants) | 8
Age, Continuous [Median (Full Range); unit: Years] | 78 [71 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 6
  More than one race | 1
  Unknown or Not Reported | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: Participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Process Outcome - Advisory Committee Members Accept Invitation
Description: Number of originally identified potential Advisory Commitee Members who accept the invitation to serve on the committee. Possible scores range from 0 to 1.
Time Frame: 1 week pre-intervention
Measure: Number; unit: Participants
Arm/Group | Experimental: occupational therapy intervention group
Number analyzed (Participants) | 1
Participants | 1

2. Primary Outcome: Process Outcome - Advisory Committee Member Participation
Description: Number of committee meetings attended by Advisory Committee Members. Possible scores range from 0 to 3.
Time Frame: Week 5 of intervention
Measure: Number; unit: Number of meetings attended
Arm/Group | Experimental: occupational therapy intervention group
Number analyzed (Participants) | 1
Number of meetings attended | 3

3. Primary Outcome: Process Outcome - Individual Activity Participation
Description: Number of individual (one-on-one) intervention activities attended by participants. Possible scores range from 0 to 6.
Time Frame: Immediately after the intervention, 6 weeks after the intervention started
Measure: Mean (Standard Deviation); unit: Number of one-on-one activities attended
Arm/Group | Experimental: occupational therapy intervention group
Number analyzed (Participants) | 8
Number of one-on-one activities attended | 5.8 (0.4)

4. Primary Outcome: Process Outcome - Group Activity Participation
Description: Number of group intervention activities attended by participants. Possible scores range from 0 to 4.
Time Frame: Immediately after the intervention, 6 weeks after the intervention started
Measure: Mean (Standard Deviation); unit: Number of group activities attended
Arm/Group | Experimental: occupational therapy intervention group
Number analyzed (Participants) | 8
Number of group activities attended | 3.5 (0.71)

5. Primary Outcome: Process Outcome - Total Activity Participation
Description: Total number of intervention activities attended by participants (individual and group). Possible scores range from 0 to 10.
Time Frame: Immediately after the intervention, 6 weeks after the intervention started
Measure: Mean (Standard Deviation); unit: # of intervention activities attended
Arm/Group | Experimental: occupational therapy intervention group
Number analyzed (Participants) | 8
# of intervention activities attended | 9.38 (0.99)

6. Primary Outcome: Process Outcome - Number Acitivites Via Zoom
Description: Number of activities attended via zoom as opposed to calling in by telephone. Possible scores range from 0 to 10.
Time Frame: Immediately after the intervention, 6 weeks after the intervention started
Measure: Mean (Standard Deviation); unit: Number of activities attended on Zoom
Arm/Group | Experimental: occupational therapy intervention group
Number analyzed (Participants) | 8
Number of activities attended on Zoom | 9.38 (0.99)

7. Secondary Outcome: Change in Self-reported Physical Activity
Description: Modified Community Health Activities Model Program questionnaire. This includes 16 questions/items that measure the number of times and the frequency of each activity engaged in during a typical week in the past month. The response scale for each of the 16 items ranges from 1=less than 1 hour to 6=9 or more hours. On this scale, higher values represent a better outcome. A total self-reported physical activity score is calculated by averaging the score of all 16 items. The range for the total score also ranges from 1 to 6. Change will be measured by creating a difference score between the pre and post intervention total scores. Positive change scores represent a better outcome, i.e., an increase in self-reported physical activity.
Time Frame: 1 week pre and 1 week post the 6-week intervention
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | Experimental: occupational therapy intervention group
Number analyzed (Participants) | 8
Units on scale | 0.20 (0.45)

8. Secondary Outcome: Change in Perceived Barriers to Physical Activity
Description: This includes 17 questions/items that measure the degree to which specific things make it more difficult for participants to engage in 30 minutes of moderate intensity physical activity on 5 or more days a week. The response scale for each of the 17 items ranges from 1=not at all more difficult to 4=much more difficult. On this scale, lower values represent a better outcome. A total perceived barriers to physical activity score is calculated by averaging the score of all 17 items. The range for the total score also ranges from 1 to 4. Change will be measured by creating a difference score between the pre and post intervention total scores. Negative change scores represent a better outcome, i.e., a decrease in perceived barriers to physical activity.
Time Frame: 1 week pre and 1 week post the 6-week intervention
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Experimental: occupational therapy intervention group
Number analyzed (Participants) | 8
Units on a scale | -0.05 (0.16)

9. Secondary Outcome: Change in Pain Interference
Description: This includes 8 questions/items that measure how much pain interferes with daily activities. The response scale for each the 8 items ranges from 1=not at all to 5=very much. On this scale, lower values represent a better outcome. A total pain interference score is calculated by averaging the score of all 8 items. The range for the total score also ranges from 1 to 5. Change will be measured by creating a difference score between the pre and post intervention total scores. Negative change scores represent a better outcome, i.e., a decrease in pain interference.
Time Frame: 1 week pre and 1 week post the 6-week intervention
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Experimental: occupational therapy intervention group
Number analyzed (Participants) | 8
Units on a scale | -0.43 (0.46)

10. Secondary Outcome: Change in Pain Intensity
Description: This includes one question about how participants rate their pain on average using a scale ranging from 0=no pain to 10=the worst imaginable pain. Change will be measured by creating a difference score between the pre and post intervention scores.
Time Frame: 1 week pre and 1 week post the 6-week intervention
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Experimental: occupational therapy intervention group
Number analyzed (Participants) | 8
Units on a scale | -1.20 (1.79)

11. Secondary Outcome: Change in Physical Function Difficulty
Description: This includes a modified version of the National Health and Aging Trends Study disability and functioning measure. The measure includes 11 questions/items assessing difficulty performing self-care, mobility, and household activities. The response scale for each of the 11 items asking about difficulty doing these activities ranges from 1=none to 4=a lot. On this scale, lower values represent a better outcome. A total physical function difficulty score is calculated by averaging the score of all 11 items. The range for the total score also ranges from 1 to 4. Change will be measured by creating a difference score between the pre and post intervention total scores. Negative change scores represent a better outcome, i.e., a decrease in physical function difficulty.
Time Frame: 1 week pre and 1 week post the 6-week intervention
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Experimental: occupational therapy intervention group
Number analyzed (Participants) | 8
Units on a scale | 0.25 (0.40)

12. Secondary Outcome: Change in Self-efficacy in Activity
Description: This includes 10 questions/items that measure participants' confidence in doing a number of activities that will be discussed during the intervention. The response scale for each of the 10 items ranges from 1=not confident at all to 5=completely confident. On this scale, higher values represent a better outcome. A total self-efficacy in activity score is calculated by averaging the score of all 10 items. The range for the total score also ranges from 1 to 5. Change will be measured by creating a difference score between the pre and post intervention total scores. Positive change scores represent a better outcome, i.e., an increase in self-efficacy in activity.
Time Frame: 1 week pre and 1 week post the 6-week intervention
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Experimental: occupational therapy intervention group
Number analyzed (Participants) | 8
Units on a scale | -0.10 (0.51)

13. Secondary Outcome: Change in Percentage of Other Participants Known
Description: This will include a measure of the percentage of other participants each participant reports knowing. Possible scores range from 0 to 100. Change will be measured by creating a difference score between the pre and post intervention scores.
Time Frame: 1 week pre and 1 week post the 6-week intervention
Measure: Mean (Standard Deviation); unit: Percentage of other participants known
Arm/Group | Experimental: occupational therapy intervention group
Number analyzed (Participants) | 8
Percentage of other participants known | 50 (35)

14. Secondary Outcome: Change in Respect Level of Other Participants
Description: This will include a measure of how much respect on average participants have for the other participants that they report knowing. This question will be asked on a scale ranging from 1=respect them very much to 5=don't respect them at all. Change will be measured by creating a difference score between the pre and post intervention scores.
Time Frame: 1 week pre and 1 week post the 6-week intervention
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Experimental: occupational therapy intervention group
Number analyzed (Participants) | 8
Units on a scale | 0.37 (0.28)

15. Secondary Outcome: Change in Sedentary Behavior
Description: Participants will be asked to wear an accelerometer for 7 days following participation in pre- and post intervention interviews. Data from the accelerometers will be used to quantify the average amount of time that participants were sedentary per day over the 7 days. Change will be measured by creating a difference score between the pre and post intervention scores.
Time Frame: 1 week pre and 1 week post the 6-week intervention
Measure: Mean (Standard Deviation); unit: Minutes per day
Arm/Group | Experimental: occupational therapy intervention group
Number analyzed (Participants) | 8
Minutes per day | 46.45 (116.36)

16. Secondary Outcome: Change in Number of Steps
Description: Participants will be asked to wear an accelerometer for 7 days following participation in pre- and post intervention interviews. Data from the accelerometers will be used to quantify the average number of steps taken per day over the 7 days. Change will be measured by creating a difference score between the pre and post intervention scores.
Time Frame: 1 week pre and 1 week post the 6-week intervention
Measure: Mean (Standard Deviation); unit: Accelerometer step count per day
Arm/Group | Experimental: occupational therapy intervention group
Number analyzed (Participants) | 8
Accelerometer step count per day | -85.5 (834.52)

ADVERSE EVENTS:
Time Frame: 10 weeks
Description: Systematic collection done by regular investigator assessment; weekly check-in intervention meetings with an occupational therapist, where adverse events were asked about and recorded
Groups:
- Experimental: occupational therapy intervention group: Behavioral: Tele-Video to Improve Daily Activity Participants will be asked to meet individually with an Occupational Therapist (OT) via Zoom to assess activity performance, establish short-term activity goals, and outline an individualized home exercise program. Participants will also be asked to participate in 4 weekly one hour group sessions via Zoom that will include: 1) education; 2) OT facilitated discussion; and 3) activity demonstration, engagement and feedback. The following topics will be covered: mobility, physical activity, pain management, and energy conservation. Participants will be asked to meet individually with the OT via Zoom for 15-20 minutes weekly to answer questions. At the end, participants will be asked to again meet individually with the OT via Zoom to re-assess activity performance and revisit short-term activity goals and the individualized home exercise program. Advisory Committee Members will be asked to make note of intervention activities during their regular interactions with other participants.
Arm/Group | Experimental: occupational therapy intervention group
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 4/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: occupational therapy intervention group (N=8)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Dizziness (Vascular disorders) | 1 (1) — Related
Fall (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated
Skin irritation (Skin and subcutaneous tissue disorders) | 1 (1) — Related, from Tegaderm
Emotional distress (Psychiatric disorders) | 1 (1) — Unrelated
Car accident (Injury, poisoning and procedural complications) | 1 (1) — Unrelated

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-09-19): https://cdn.clinicaltrials.gov/large-docs/64/NCT06007664/Prot_SAP_001.pdf
  • Informed Consent Form (2023-06-19): https://cdn.clinicaltrials.gov/large-docs/64/NCT06007664/ICF_000.pdf